CLINICAL TRIAL: NCT01578954
Title: LCCC 1111: An Open-Label Dose-Finding Study of Lenalidomide as Reinduction/ Consolidation Followed by Lenalidomide Maintenance Therapy for Adults ≥ 60 Years of Age With Acute Myeloid Leukemia (AML) in Partial or Complete Response Following Conventional Induction Therapy
Brief Title: Lenalidomide as Consolidation and Maintenance in Adults >/= 60 Years of Age With AML Following Standard Induction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1111; 12-0040 (Other: UNC - Biomedical IRB)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug (Experimental): Lenalidomide (25, 35, or 50 mg induction/10mg maintenance)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Reinduction/Consolidation - dose escalation of lenalidomide: Level 1 - 25mg, Level 2 - 35mg, Level 3 - 50mg, PO, QD, 28 days.
  Maintenance Lenalidomide - 10mg, PO, QD, continuous dosing, 12 months
  Other Names: Revlimid

SUMMARY:
The purpose of this research study is to test the safety of the study drug, lenalidomide, at different dose levels in people diagnosed with acute myeloid leukemia (AML) who have finished standard induction therapy and have had a partial or complete response to induction therapy. The investigators want to find out what effects (for example, side effects) the study drug, lenalidomide, has on people and their leukemia. The investigators also want to see if additional treatment (maintenance therapy) with lenalidomide will keep the leukemia from relapsing (coming back).

DETAILED DESCRIPTION:
This study is a single-arm, open-label phase Ib clinical trial testing the hypothesis that the daily use of lenalidomide will be safe and tolerable as evidenced by the rate of dose-limiting toxicity (DLT) seen during one month of reinduction/consolidation in older (≥ 60 years of age) acute myeloid leukemia (AML) patients treated after one cycle of conventional, anthracycline-based induction. (Re-induction is the prescribed lenalidomide therapy given to patients who are in partial remission/response post induction while consolidation is the same prescribed lenalidomide therapy post induction given to patients who are in complete remission).

Dose escalation will take place within cohorts during the 28-day re-induction/ consolidation lenalidomide treatment at the University of North Carolina at Chapel Hill. After re-induction/consolidation, patients who harbor ≥ 5% peripheral blood or bone marrow myeloblasts will be removed from protocol therapy. Patients who have <5% peripheral blood or bone marrow myeloblasts after consolidation therapy will be allowed to continue to maintenance therapy: lenalidomide 10 mg/day continuously for up to 12 months. Up to 26 patients will be enrolled.

This trial includes a Geriatric Assessment (GA) of each enrolled patient at baseline and serially across the trial. The investigators also plan to study natural killer (NK) cell phenotype and cytolytic function in patients at various intervals across the study (baseline, post re-induction/consolidation, and during maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥60 years of age with AML

  * Patients with therapy-related myeloid neoplasms are allowed
  * Patients with AML that has evolved from an antecedent hematologic disorder are allowed
  * Patients will be eligible regardless of their ultimate plans or candidacy for allogeneic stem cell transplant
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP; see definition below) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for re-induction/consolidation (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.

  * A FCBP is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix C: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Patients must have been treated with 1-2 courses of intensive therapy as first therapy for AML, commonly described as induction. These therapies should include cytarabine at a dose ≥700 mg/m2 in combination with an anthracycline or anthracenedione (≥ 135 mg/m2 of daunorubicin, 36 mg/m2 of idarubicin or 40 mg/m2 of mitoxantrone)
* Patients must be in morphologic complete response (CR), complete response with incomplete hematologic recovery (CRi) or partial response (PR) by international working group criteria post induction therapy (see Appendix A). Patients in PR who have undergone only one course of intensive induction therapy will be eligible only if one or more of the following criteria are met:

  * Patient preference to forgo further intensive induction therapy in favor of low- or intermediate-intensity therapy
  * Patients are deemed unlikely to benefit from additional anthracycline-cytarabine induction therapies for any of the following reasons:

    * Therapy-related AML
    * Prior myelodysplastic syndrome or myeloproliferative neoplasm
    * The presence of cytogenetic or molecular genetic features place patient in the Intermediate-I, Intermediate -II or Adverse genetic group as defined by the European LeukemiaNet
  * Patients who have experienced one or more CTCAE v4.0 grade 3-4 treatment-related non-hematologic toxicity within 30 days of beginning the first course of induction therapy.
* Patients must have recovered from all infectious and non-hematologic toxicities from prior chemotherapy to ≤ CTCAE grade 1 or baseline prior to study enrollment.
* Adequate renal and hepatic functions as indicated by the following:

  * Renal function assessed by calculated creatinine clearance (CrCl) must be >/= 60ml/min by Cockcroft-Gault formula (
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST/ALT ≤ 2.5 x ULN
* Patients in CRi must have evidence of hematologic recovery after prior therapy to at least:

  * Absolute neutrophils ≥ 0.8 x 109/L
  * Platelets ≥ 75 x 109/L
  * Independent of red blood cell transfusions
* ECOG performance status 0-2

Exclusion Criteria:

* Prior treatment with lenalidomide
* Known hypersensitivity to thalidomide
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* The diagnosis of AML-M3 (acute promyelocytic leukemia) characterized by translocations involving the retinoic acid receptor-alpha (RAR-alpha) gene.
* Use of investigational agents within 2 weeks or any anticancer therapy within 2 weeks before study entry; the patient must have recovered from all acute toxicities from any previous therapy.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive because of hepatitis B vaccine are eligible.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Have currently active gastrointestinal disease, or prior surgery that may affect the ability of the patient to absorb oral lenalidomide

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06-28 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

PRIMARY OUTCOMES:
Determine the rate of dose limiting toxicities. | 28 days

SECONDARY OUTCOMES:
Frequency of toxicity | 28 days
  Number of adverse events that occur during induction/consolidation.
Duration of toxicity | 28 days
  Duration is measured by the length of time of a toxicity to resolve or return to baseline that occur during induction.
Frequency of toxicity | 12 months
  Frequency will be measured as the number of individual toxicities that occur during maintenance.
Response rates | 12 months
  Response is based on the International Working Group to standardize response in AML.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Foster, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Woods JD, Zeidner JF, Van Deventer HW, Jamieson K, Matson M, Zhang J, Pulley W, Brenizer T, Muss H, Nyrop KA, Vohra SN, Deal AM, Ivanova A, Foster MC. Phase Ib trial of lenalidomide as post-remission therapy for older adults with acute myeloid leukemia: Safety and longitudinal assessment of geriatric functional domains. J Geriatr Oncol. 2022 May;13(4):499-504. doi: 10.1016/j.jgo.2021.11.015. Epub 2021 Dec 23. PMID 34955443
- See also: Lineberger Comprehensive Cancer Center Website — http://unclineberger.org/